CLINICAL TRIAL: NCT05871944
Title: Effectiveness of Kaltenborn End Range Joint Mobilization Technique and Post Facilitation Stretch in Shoulder Impingement Syndrome
Brief Title: Effectiveness of Kaltenborn End Range Joint Mobilization Technique and Post FacilitationStretch in Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Collaborators: Al Nafees Medical Hospital, Islamabad (Unknown); National Institute of Rehabilitation Medicine, Islamabad, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 341
Record Dates: First submitted 2023-05-13; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Two groups will be formed. one group will receive joint mobilization technique and other will get post facilitation stretch technique
Who Masked: Participant
Masking Description: This will be single blind randomized control clinical trail in which just participant will be unware about which group he/she is included
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): kalternborn joint mobilization techniques will be administered for total of 8 weeks at the rate of 2 session per week.
  Interventions: Other: KAlternborn Joint Mobilization
- experimental group (Experimental): Post stretch facilitation technique will be administered for total of 8 weeks at the rate of 2 session per week.
  Interventions: Other: Post stretch Facilitation Technique

INTERVENTIONS:
Other: KAlternborn Joint Mobilization — This is a join mobilization technique to reduce the joint stiffness and help in improving joint range of motion
  Arms: control group
Other: Post stretch Facilitation Technique — This is a PNF techniques used to relax the muscles and help in getting more free range of restricted joint
  Arms: experimental group

SUMMARY:
This study is a experimental one to observe the efficacy of joint mobilization and post facilitation techniques in shoulder impingement syndrome

DETAILED DESCRIPTION:
his study is a experimental one to observe the efficacy of Kalternborn end range joint mobilization and post facilitation techniques in shoulder impingement syndrome. Goniometer, shoulder disability index will be the tool used for evaluation

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age 25 to 45
* Diagnosed Rotator cuff impingement from ortho, neuro and musculoskeletal department
* Hawkin kennedy test positive
* Neer's test positive
* Jobe's test positive

Exclusion Criteria:

* Cervical spine disorder
* Fractures
* Major upper limb surgery
* Tumor or wound
* Diagnosed acromial malformations

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Goniometer | 4 weeks
  This is a instrument designed to evaluate the joint range of motion. Greater ranges mean more mobility of joint and less means more restriction
Shoulder Pain and Disability Index | 4 weeks
  Used to assess the patients level of pain and the ADLs which are affected. O score means no dysfuction of joint and higer score means more dysfuction

CONTACTS AND LOCATIONS:
Locations (1):
- Al Nafees Medical Hospital, Islamabd, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Have not decided yet about this.